CLINICAL TRIAL: NCT00743977
Title: 2 Treatment, 2 Period, Randomized, Single Blinded, Crossover Bioequivalence of Phenazopyridine HCl in 24 Healthy Volunteers
Brief Title: Bioequivalence of Phenazopyridine HCl in Healthy Volunteers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universal Enterprises (Industry)
Responsible Party: Head of Clinical Research, Universal Research Group
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: URG/STEROP/001
Record Dates: First submitted 2008-08-28; First posted 2008-08-29 (Estimated); Last update posted 2008-08-29 (Estimated); Status verified 2008-08

CONDITIONS: Human Volunteers
MeSH Terms: interventions — Phenazopyridine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator)
  Interventions: Drug: Phenazopyridine HCl
- B (Experimental)
  Interventions: Drug: Phenazopyridine HCl

INTERVENTIONS:
Drug: Phenazopyridine HCl — 100mg tablet in fasting state
  Other Names: Pyridium

SUMMARY:
The present study aims at comparing the pharmacokinetics of the original formulation of phenazopyridine and a same generic product.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects aged 18 to 55 (Male & Female)
* Physically and mentally healthy subjects as confirmed by an interview, medical history, clinical examination, laboratory tests
* Informed consent signed by the subject
* The subject is co-operative and available for the entire study
* Not pregnant or nursing
* Normal renal and hepatic function

Exclusion Criteria:

* Evidence in the subject medical history or in the medical examination of any clinically significant hepatic, renal, gastrointestinal, cardiovascular, pulmonary, hematological or other significant acute or chronic abnormalities which might influence either the safety of the subject or the absorption, distribution, metabolism or excretion of the active agent under investigation
* Hypersensitivity to subject drug, atopic eczema or allergic bronchial asthma
* Evidence of hypertension (blood pressure after 3 minutes sitting>160/95 mm Hg)
* Evidence of chronic or acute infectious diseases;
* History or evidence of malignant tumors;
* Evidence of hyperuricaemia, elevated serum uric acid (>8.0 mg/dl)
* Hepatic or renal impairment; elevated serum creatinine (>1.4 mg/dl)
* Planned vaccination during the time course of the study
* Adherence to a diet (i.e, vegetarian) or life style (incl. extreme sports) that might interfere with the investigation
* Laboratory test results outside the tolerance values as laid down by the study centre, which may be an evidence of disease. Positive result of HIV1/2, HCV antibody or HBs antigen testing
* Regular use of any medication within four weeks prior to commencement of the study (self-medication or prescription)
* Single use of any medication (including OTC) that are not expressively permitted within two weeks prior to start of the study
* Abuse of alcohol, caffeine or tobacco (equivalent to more than 10 cigarettes a day)
* Drug addiction
* Participation in a clinical investigation or blood donation of more than 250 ml within the past eight weeks or blood donation of less than 250 ml within the past 4 week
* Subjects who are known or suspected

  * not to comply with the study directives
  * not to be reliable or trustworthy
  * not to be capable of understanding and evaluating the information given to them as part of the formal information policy (informed consent),in particular regarding the risks and discomfort to which they would agree to be exposed.
  * to be in such a precarious financial situation that they no longer weigh up the possible risks of their participation and the unpleasantness they may be involved in.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2008-08; Primary Completion 2008-11 (Estimated)

PRIMARY OUTCOMES:
The primary outcome of the study will be to determine the bioequivalence of both the formulations of phenazopyridine | regular intervals after drug dosing

CONTACTS AND LOCATIONS:
Overall Officials: Waqar H. Kazmi, M.D, M.S., Principal Investigator
Locations (1):
- Health Care Hospital, Karachi, Pakistan